CLINICAL TRIAL: NCT00127192
Title: Sitagliptin (MK0431) Late Phase II Double-Blind Dose-Response Study - Type 2 Diabetes Mellitus
Brief Title: A Study of an Investigational Drug Sitagliptin for Type 2 Diabetes Mellitus (0431-044)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-044; MK0431-044; 2005_037
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Placebo Comparator): Placebo QD 12-week
  Interventions: Drug: Comparator: placebo (unspecified)
- 2 (Experimental): 25 mg QD 12-week
  Interventions: Drug: sitagliptin phosphate
- 3 (Experimental): 50 mg QD 12-week
  Interventions: Drug: sitagliptin phosphate
- 4 (Experimental): 100 mg QD 12-week
  Interventions: Drug: sitagliptin phosphate
- 5 (Experimental): 200 mg QD 12-week
  Interventions: Drug: sitagliptin phosphate

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin phosphate 25 mg, 50 mg, 100 mg QD, or 200 mg QD 12-weeks.
  Other Names: MK0431
  Arms: 2; 3; 4; 5
Drug: Comparator: placebo (unspecified) — placebo QD 12-weeks
  Arms: 1

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of an investigational drug in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus

Exclusion Criteria:

* Patients with type 1 diabetes mellitus

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Iwamoto Y, Taniguchi T, Nonaka K, Okamoto T, Okuyama K, Arjona Ferreira JC, Amatruda J. Dose-ranging efficacy of sitagliptin, a dipeptidyl peptidase-4 inhibitor, in Japanese patients with type 2 diabetes mellitus. Endocr J. 2010;57(5):383-94. doi: 10.1507/endocrj.k09e-272. Epub 2010 Mar 24. PMID 20332588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase II.
  First patient in: 11 July 2005. Last patient, last visit: 8 March 2006.
  The study was conducted at 97 centers in Japan.
Pre-assignment Details: Patients 20-75 years of age with type 2 diabetes mellitus and inadequate glycemic control (HbA1c ≥6.5% and <10% at Week -2) were eligible for randomization following at least 8 weeks of diet/exercise and antihyperglycemic agent (AHA) wash-off (for patients previously on an AHA), including a 2-week placebo run-in.
Groups:
- Sitagliptin 25 mg QD: The Sitagliptin 25 mg group includes data from all patients randomized to receive treatment with sitagliptin 25 mg orally once daily (QD=once daily).
- Sitagliptin 50 mg QD: The Sitagliptin 50 mg group includes data from all patients randomized to receive treatment with sitagliptin 50 mg orally once daily (QD=once daily).
- Sitagliptin 100 mg QD: The Sitagliptin 100 mg group includes data from all patients randomized to receive treatment with sitagliptin 100 mg orally once daily (QD=once daily).
- Sitagliptin 200 mg QD: The Sitagliptin 200 mg group includes data from all patients randomized to receive treatment with sitagliptin 200 mg orally once daily (QD=once daily).
- Placebo: The Placebo group includes data from all patients randomized to receive treatment with matching placebo orally once daily.
Period: Overall Study
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Started | 80 (Study enrolled slightly more than the target of N=70) | 72 (Study enrolled slightly more than the target of N=70) | 70 (Study enrolled as per the target of N=70) | 68 (Study enrolled slightly less than the target of N=70) | 73 (Study enrolled slightly more than the target of N=70)
Completed | 77 | 71 | 68 | 67 | 68
Not Completed | 3 | 1 | 2 | 1 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 3
Not completed — Adverse event in pre-treatment period | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo | Total
Number analyzed (Participants) | 80 | 72 | 70 | 68 | 73 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (7.9) | 60.2 (9.4) | 58.3 (9.5) | 60.6 (7.7) | 60.2 (8.0) | 59.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 34 | 28 | 23 | 139
  Male | 51 | 47 | 36 | 40 | 50 | 224
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 145.7 (37.6) | 144.3 (29.0) | 142.6 (31.8) | 148.4 (33.3) | 156.5 (35.1) | 147.5 (33.8)
Glycosylated albumin [Mean (Standard Deviation); unit: percent] | 21.5 (3.9) | 22.0 (4.2) | 21.9 (4.5) | 21.9 (3.9) | 23.7 (4.5) | 22.2 (4.3)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.5 (0.8) | 7.6 (0.8) | 7.6 (0.8) | 7.7 (0.8) | 7.7 (0.9) | 7.6 (0.8)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Glycosylated Albumin at Week 12
Description: Change from baseline at Week 12 is defined as Week 12 minus Week 0.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. For FAS patients with no data at Week 12, the last non-baseline observed measurement was carried forward to Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Number analyzed (Participants) | 80 | 72 | 70 | 68 | 73
Percent | -1.9 [-2.4 to 1.5] | -2.6 [-3.1 to 2.2] | -2.6 [-3.0 to 2.1] | -2.9 [-3.4 to 2.5] | 0.7 [0.2 to 1.1]
Statistical Analysis 1: Comparison: Sitagliptin 200 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — Multiplicity among pairwise comparisons of sitagliptin groups against placebo was adjusted by Bonferroni method in post-hoc manner; ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline was used for pairwise comparison; Least-squares Mean Difference = -3.6, 95% CI [-4.3 to -3.0] — ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline was used to estimate difference of two groups and its 95% confidence interval
Statistical Analysis 2: Comparison: Sitagliptin 100 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -3.2, 95% CI [-3.9 to -2.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -3.3, 95% CI [-3.9 to -2.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sitagliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -2.6, 95% CI [-3.2 to -2.0] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Number analyzed (Participants) | 80 | 72 | 70 | 68 | 73
Percent | -0.41 [-0.52 to 0.29] | -0.71 [-0.83 to 0.59] | -0.69 [-0.81 to 0.56] | -0.76 [-0.89 to 0.64] | 0.28 [0.16 to 0.40]
Statistical Analysis 1: Comparison: Sitagliptin 25 mg QD vs Sitagliptin 50 mg QD vs Sitagliptin 100 mg QD vs Sitagliptin 200 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Tukeys linear trend test based on ANCOVA; Linear contrast including all groups was tested using ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline
Statistical Analysis 2: Comparison: Sitagliptin 200 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — No multiplicity adjustment was done between trend test of primary analysis and pairwise comparisons, but the multiplicity among pairwise comparisons of sitagliptin groups against placebo was adjusted by Bonferroni method in post-hoc manner; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -1.04, 95% CI [-1.21 to -0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — No multiplicity adjustment was done between trend test of primary analysis and pairwise comparisons, the multiplicity among pairwise comparisons of sitagliptin groups against placebo was adjusted by Bonferroni method in post-hoc manner; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -0.96, 95% CI [-1.14 to -0.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sitagliptin 50 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -0.99, 95% CI [-1.16 to -0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Sitagliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -0.69, 95% CI [-0.85 to -0.52] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: Change from baseline at Week 12 is defined as Week 12 minus Week 0.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Number analyzed (Participants) | 80 | 72 | 70 | 68 | 73
mg/dL | -9.6 [-14.0 to 5.3] | -11.4 [-16.0 to 6.8] | -14.6 [-19.2 to 9.9] | -16.9 [-21.6 to 12.1] | 6.3 [1.7 to 10.9]
Statistical Analysis 1: Comparison: Sitagliptin 200 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -23.2, 95% CI [-29.8 to -16.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -20.8, 95% CI [-27.4 to -14.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -17.7, 95% CI [-24.2 to -11.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sitagliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -15.9, 95% CI [-22.3 to -9.6] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Reported overdoses, regardless of association with reported adverse events, were considered as serious adverse events in this study. The patients for whom the event of overdose was reported had no concomitant AEs with the overdose.
Arm/Group | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 0 | 2 | 0
Other Adverse Events (participants affected / at risk) | 31 | 25 | 32 | 20 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Angina pectoris (Cardiac disorders) | 0/80 | 1/72 | 0/70 | 0/68 | 0/73
Cardiac failure chronic (Cardiac disorders) | 0/80 | 0/72 | 0/70 | 1/68 | 0/73
Hypertensive heart disease (Cardiac disorders) | 0/80 | 0/72 | 0/70 | 1/68 | 0/73
Myocardial ischaemia (Cardiac disorders) | 0/80 | 0/72 | 0/70 | 1/68 | 0/73
Overdose (Injury, poisoning and procedural complications) | 0/80 | 0/72 | 0/70 | 1/68 | 0/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 25 mg QD | Sitagliptin 50 mg QD | Sitagliptin 100 mg QD | Sitagliptin 200 mg QD | Placebo
Constipation (Gastrointestinal disorders) | 6/80 | 2/72 | 3/70 | 1/68 | 3/73
Nasopharyngitis (Infections and infestations) | 16/80 | 16/72 | 23/70 | 12/68 | 17/73
Pharyngitis (Infections and infestations) | 0/80 | 2/72 | 4/70 | 2/68 | 0/73
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3/80 | 3/72 | 2/70 | 4/68 | 3/73
Headache (Nervous system disorders) | 0/80 | 1/72 | 0/70 | 1/68 | 5/73
Alanine aminotransferase increased (Investigations) | 0/80 | 4/72 | 0/70 | 0/68 | 1/73
Blood creatine phosphokinase increased (Investigations) | 7/80 | 2/72 | 1/70 | 1/68 | 2/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.